CLINICAL TRIAL: NCT01819376
Title: Use of Facebook as a Motivating Factor in a Weight-reduction Program for Obese and Overweight Adolescents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TecSalud Investigación Clínica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ADOBFB
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Overweight; Adolescents; Teenagers; Facebook; Social Networks
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Facebook updates (Experimental): The experimental group will be encouraged to update their Facebook status regarding healthy lifestyle decisions at least once a day.
  Interventions: Other: Facebook Status Update
- Control: No Facebook (No Intervention): This group will be encouraged not to share their healthy lifestyle decisions on Facebook.

INTERVENTIONS:
Other: Facebook Status Update
  Arms: Intervention: Facebook updates

SUMMARY:
The purpose of this study is to determine if Facebook can be used as a motivating factor for obese or overweight adolescents in a weight-reduction program.

DETAILED DESCRIPTION:
This study is a randomized controlled trial. There will be two randomly assigned groups of obese or overweight adolescents (WHO definition). Both groups will be enrolled in a 12 week weight reduction program which includes personal nutritional evaluation and food plan and exercise routine. Follow-up appointments will be held every 3 weeks. One group will be encouraged to update their Facebook status at least once a day, regarding their healthy lifestyle changes (exercise routine, healthy food choice, "checking-in" at the wellness center, kilograms lost, etc). The control group will be asked not to share information about their program on Facebook for 12 weeks. Facebook follow-up will be held by the investigators on the study's Facebook account. Teenagers will be thoroughly explained on how to set the account to a limited profile if they want to. At the end of the program both groups will be compared regarding weight loss and mean BMI.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 13 and 19 years old.
* Obese or overweight according to the IOTF.
* No physical or medical impediment for performing physical activity.
* No risk for eating disorders (SCOFF questionnaire).
* Report less than 20 minutes of physical activity per day.
* Have an active Facebook account and use it more than 20 minutes per day.
* Low-risk in the Gatehouse Bullying Scale.

Exclusion Criteria:

* Physical or medical impediment for performing physical activity.
* Answer "yes" at least twice on the SCOFF questionnaire.
* Report more than 20 minutes of exercise per day.
* Not having an active Facebook account or using it less than 20 minutes per day.
* "High Risk" on the Gatehouse Bullying Scale.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
BMI | 12 weeks
  Body Mass Index

SECONDARY OUTCOMES:
Positive Feedback | 12 weeks
  Positive feedback ("likes", positive comments) will be evaluated and related to BMI reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Bienestar Integral, Monterrey, Nuevo León, Mexico